CLINICAL TRIAL: NCT02503306
Title: Clinical Trial on Efficacy and Tolerability of Two Different Single Doses of Avanafil in Russia
Brief Title: Efficacy and Tolerability Study of Avanafil in Russia
Acronym: CEDAR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AVANAL07163; U1111-1167-6889 (Other: UTN)
Record Dates: First submitted 2015-07-17; First posted 2015-07-20 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Sexual Function and Fertility Disorders NEC-Erectile Dysfunction
MeSH Terms: interventions — avanafil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Avanafil dose 1 (Experimental): Administered 30 minutes prior to initiation of sexual activity for a duration of 8 weeks to use no more than one dose in any 24-hour period
  Interventions: Drug: AVANAFIL
- Avanafil dose 2 (Experimental): Administered 30 minutes prior to initiation of sexual activity for a duration of 8 weeks to use no more than one dose in any 24-hour period
  Interventions: Drug: AVANAFIL
- Placebo (Placebo Comparator): Administered 30 minutes prior to initiation of sexual activity for a duration of 8 weeks to use no more than one dose in any 24-hour period
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: AVANAFIL — Pharmaceutical form:tablets Route of administration: oral
  Arms: Avanafil dose 1; Avanafil dose 2
Drug: placebo — Pharmaceutical form:tablets Route of administration: oral
  Arms: Placebo

SUMMARY:
Primary Objective:

o To assess the change in percent of sexual attempts in which subjects are able to maintain an erection of sufficient duration to have successful intercourse between the run-in period and treatment period:

* The change in percent of sexual attempts in which subjects are able to insert the penis into the partner's vagina.
* The change in score on the erectile function (EF) domain of the International Index of Erectile Function (IIEF) questionnaire.

Secondary Objective:

o To evaluate the safety and tolerability of avanafil in patients with erectile dysfunction (ED).

DETAILED DESCRIPTION:
The total study duration per patient will be up to 12 weeks, consisting of an 8-week treatment period and a 4-week run-in period.

ELIGIBILITY:
Inclusion criteria:

* Male subjects, age ≥18 years.
* Minimum 6-month history of mild to severe erectile dysfunction prior to the enrollment into the study.
* Subject is in a monogamous, heterosexual relationship for at least 3 months prior to the enrollment into the study.
* Subject agrees to make at least 4 sexual intercourse attempts per month.
* Subject is willing and able to provide informed consent.

Exclusion criteria:

* Allergy or hypersensitivity to avanafil, sildenafil, vardenafil, tadalafil, or any of the components of these drug products.
* History of dose-limiting adverse effects during therapy with a phosphodiesterase-5 (PDE5) inhibitor or history of consistent treatment failure with other PDE5 inhibitors for therapy of ED.
* Current or expected use of organic nitrates at any time during the study.
* Previous or current (including while on treatment) antiandrogen therapy.
* Use of ketoconazole, erythromycin, cimetidine, or any other prescription or over-the-counter drugs known to inhibit the activity of cytochrome P450 (CYP) 3A4 within 28 days prior to randomization or at any time during this study.
* Androgen replacement therapy that has not been stable for at least 3 months.
* Erectile dysfunction as a result of spinal cord injury or radical prostatectomy.
* Untreated hypogonadism or serum total testosterone <325 ng/dL (early morning collection).
* History of or predisposition to priapism (such as sickle cell disease, blood dyscrasias, or multiple myeloma).
* Uncontrolled hypertension as evidenced by systolic blood pressure >170 mmHg or diastolic blood pressure >100 mmHg at screening.
* Hypotension as evidenced by systolic blood pressure <90 mmHg or diastolic blood pressure <50 mmHg at screening.
* Orthostatic hypotension as evidenced by reduction of 20 mmHg or more in systolic blood pressure, reduction of 10 mmHg or more in diastolic blood pressure, or evidence of cerebral hypoperfusion upon standing from a seated position.
* Clinically evident penile lesions, abrasions, anatomical deformities such as penile fibrosis, Peyronie's disease, urinary tract or bladder infection, or sexually transmissible disease that the Investigator deems to be clinically significant.
* History of drug, alcohol, or substance abuse within 12 months of entry.
* Partners who are <18 years of age, who are nursing, who are known to be pregnant at screening, who wish to become pregnant during the study period, who have dyspareunia, and/or any other gynecologic problems or major medical conditions that would limit participation in sexual intercourse.
* Evidence of any clinically significant medical, psychiatric, social, or other condition by history, physical examination, or laboratory studies that, in the opinion of the Investigator, would contraindicate the administration of study medication, affect compliance, interfere with study evaluations, limit study participation, contraindicate sexual activity, or confound the interpretation of study results.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2015-07; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Change in the percentage of sexual attempts in which subjects are able to maintain an erection of sufficient duration to have successful intercourse | 12 weeks
Change in the percentage of sexual attempts in which subjects are able to insert the penis into the partner's vagina | 8 weeks
Change from baseline in EF score | baseline and 8 weeks

SECONDARY OUTCOMES:
Change from baseline in IIEF-EF risk scores | baseline and 8 weeks
Proportion of patients with adverse events | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Moscow, Russia